CLINICAL TRIAL: NCT00003582
Title: Phase I/II Study to Evaluate Combined Hyperfractionated Radiation Therapy and 5-Fluorouracil, Cisplatin and Paclitaxel (Taxol) and Amifostine (WR 2721, Ethyol) in Stage III and IV Inoperable Head and Neck Carcinomas
Brief Title: Radiation Therapy, Combination Chemotherapy, and Amifostine in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Purpose: Treatment
Other Study IDs: 88191; SCCC-1988007 (Other: University of Miami Sylvester Comprehensive Cancer Center); ALZA-97-052-ii; BHM-98-32; NCI-V98-1474
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Carcinoma of Unknown Primary; Head and Neck Cancer
Keywords: squamous cell carcinoma of unknown primary; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Neoplasms, Unknown Primary; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Amifostine; Cisplatin; Fluorouracil; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: fluorouracil
Drug: paclitaxel
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of radiation therapy and chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy plus combination chemotherapy and amifostine in treating patients who have stage II, stage III, or stage IV head and neck cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the impact of amifostine on the acute tolerance of combined hyperfractionated radiation therapy and fluorouracil, cisplatin, and paclitaxel with amifostine, in terms of the grade and duration of acute mucositis and dermatitis, and acute hematologic tolerance in patients with stage III or IV unresectable head and neck carcinoma. II. Determine the local control and survival associated with this regimen in these patients. III. Determine the long term chronic toxic effects of this regimen in terms of swallowing dysfunction, PEG dependency, and xerostomia in these patients. IV. Determine the quality of life post therapy by assessment of speech and swallowing function in these patients. V. Determine if radiation dose escalation in patients with treatment interruption achieve an isoeffect on locoregional control. VI. Determine the safe optimal dose of paclitaxel to be combined with hyperfractionated radiation therapy, fluorouracil, cisplatin, and amifostine in these patients. VII. Determine the correlation of p53 chromosome expression on locoregional control and survival of these patients. VIII. Quantitate tumor volumetrics and correlate with stage, resectability status, and locoregional control and survival of these patients.

OUTLINE: This is a dose escalation of paclitaxel, multicenter study. Patients are stratified by performance status, stage, institution, tumor volumetrics, resectability, and p53 expression. Patients receive amifostine IV over 10 minutes on Monday of weeks 1, 5, and 9, and over 5-7 minutes Tuesday through Friday of weeks 1, 5, and 9 and Monday through Friday of weeks 2, 3, 4, 6, and 7. Within 10-15 minutes of amifostine administration, patients receive paclitaxel IV over 3 hours, cisplatin IV over 2 hours on days 1, 29, and 56, and fluorouracil IV over 72 hours on days 1-4, 29-33, and 56-60. Starting on day 2, patients receive hyperfractionated external beam radiotherapy twice daily over 6.5 weeks, following amifostine IV over 5-7 minutes Monday through Friday. Cohorts of 6-20 patients each receive escalating doses of paclitaxel. Quality of life is assessed. Patients are followed monthly for 1 year, every 2 months for 1 year, every 6 months for 3 years, and then annually thereafter until death.

PROJECTED ACCRUAL: A minimum of 36 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck, including: Stage III or IV: oral cavity, paranasal sinus, hypopharynx, oropharynx, larynx, and nasopharynx OR Unknown primary carcinoma of the head and neck with greater than N1 disease if no planned neck dissection Evaluable disease No metastases below clavicle by clinical or radiographic diagnosis All hypopharynx and nasopharynx patients with N3 disease undergo a CT scan of the chest

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Platelet count at least 130,000/mm3 WBC at least 3,400/mm3 Hemoglobin greater than 10.0 g/dL (transfusion allowed) Hepatic: Not specified Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: No active heart disease No myocardial infarction within past 6 months No uncontrolled congestive heart failure No uncontrolled angina Cardiac ejection fraction at least 50% by MUGA scan for patients under 65 without antecedent heart disease, at least 55% for patients over 65 and/or with antecedent heart disease Pulmonary: FEV greater than 60% of predicted Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the treatment field Surgery: Eligible for PEG gastrostomy Other: At least 24 hours since prior antihypertensive and diuretic medications (prior to amifostine and chemotherapy regimens)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1988-05; Primary Completion 1996-12 (Actual); Study Completion 1996-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre A. Abitbol, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- Sylvester Cancer Center, University of Miami, Miami, Florida, United States